CLINICAL TRIAL: NCT04601818
Title: Planned Semi-Elective Lung Transplantation Using 10C Cold Static Preservation: A Proof-Of-Concept Study
Brief Title: Planned Semi-Elective Lung Tx Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB202001646
Record Dates: First submitted 2020-07-16; First posted 2020-10-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: To Compare Lung Transplant Outcomes Between Study Patients and Standard Patients Who Have Already Undergone Lung Transplantation by Conventional Procedures; Lung Transplant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional arm (Experimental): During our study period, transplants with a planned recipient anesthesia starting time between 10:00pm-6:00am will be allowed to move to a 6:00-8:00am start at the earliest. To be eligible, donor lungs cross clamp time have to occur between 6pm and 4am and lungs need to be suitable for transplantation without the need for ex vivo lung evaluation. Lungs meeting criteria for direct transplantation will be transported in the usual fashion in a cooler of ice at 4oC and upon arrival to Shands UF Health they will immediately be transferred to cold static preservation at 10oC within a specific refrigerator placed in the Shands UF Health OR. The maximum preservation time from donor cold flush (cross clamp) to recipient anesthesia start should be 12 hours and the recipient procedure should not start before 6am.
  Interventions: Procedure: Experimental: Preserving of Donor Lungs
- Retrospective arm (No Intervention): Outcomes will be compared to conventional transplant patients matched by age, medical diagnosis, BMI, lung allocation score and donor type ( DCD vs. NDD) using a 1:2 matching.

INTERVENTIONS:
Procedure: Experimental: Preserving of Donor Lungs — lung transplants that have a proposed after hours start time will be delayed until 6am and the donor lungs will be preserved for no more than 12 hours at 10 degrees celsius cold static
  Arms: Interventional arm

SUMMARY:
When suitable donor lungs become available for a consented recipient, and the donor cross clamp time occurs between 6pm and 4am, the transplant procedure (anesthesia starting time) will be allowed to be moved to a 6am start or later with the lungs being preserved at 10C cold static preservation upon organ arrival to our hospital using a specific refrigerator. The maximum allowed time between donor cross clamp and recipient anesthesia initiation will be 12h.

ELIGIBILITY:
Inclusion Criteria:

* Primary lung transplantation
* Informed consent provided

Donor Inclusion: Age<70

Exclusion Criteria:

* Re-transplantation
* Multi-organ transplantation

Donor exclusion criteria:

* Age >70y
* Concerns with organ preservation technique

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of ISHLT Primary Graft Dysfunction Grade 3 at 72 hours (expected rate less than 20%) | 72 hours post op

SECONDARY OUTCOMES:
1-year survival | procedure up to 1 year post op

CONTACTS AND LOCATIONS:
Overall Officials: Mindaugas Rackauskas, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- UFHealth Shands, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No